CLINICAL TRIAL: NCT04826926
Title: Impact of Timing of Re-evaluation After Non-surgical Periodontal Therapy on Clinical Parameters and Decision-making. A Prospective Clinical Trial
Brief Title: Timing of Periodontal Re-evaluation After Non-surgical Periodontal Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UTurin02
Record Dates: First submitted 2021-03-23; First posted 2021-04-01 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-01

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non-surgical periodontal treatment NSPT (Experimental): Conventional staging debridement (CSD) according to the severity of periodontal disease in 2 to 4 appointments at day 0, 7, 14 and 21.
  Supra and subgingival scaling and polishing will be performed by the use of manual and ultrasonic instruments and oral hygiene instructions will be given. Patients will be instructed to use interdental brushes with appropriate size interdental brushes or dental floss when interdental embrasures will not allow for interdental brushing.
  Interventions: Procedure: Procedure/Surgery: Non Surgical Periodontal Therapy

INTERVENTIONS:
Procedure: Procedure/Surgery: Non Surgical Periodontal Therapy — Conventional staging debridement (CSD) according to the severity of periodontal disease in 2 to 4 appointments at day 0, 7, 14 and 21.
  Supra and subgingival scaling and polishing will be performed by the use of manual and ultrasonic instruments and oral hygiene instructions will be given. Patients will be instructed to use interdental brushes with appropriate size interdental brushes or dental floss when interdental embrasures will not allow for interdental brushing.

SUMMARY:
Literature on non surgical periodontal therapy (NSPT) shows lack of clarity in reporting information on re-evaluation timing and clinical response. If the re-evaluation was done shortly after NSPT, this is also likely to have an influence on the surgical treatment plan. The aim of this prospective clinical trial is to investigate the effect of re-evaluation timing at 1-3-6 months after NSPT in terms of pocket closure, PD reduction, comprehensive treatment plan, and costs for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Periodontitis stage III-IV
* Full-mouth plaque score (FMPS) < 25% at the 1-month re-evaluation
* Full-mouth bleeding score (FMBS) < 25% at the 1-month re-evaluation
* Signed informed consent

Exclusion criteria

* Age < 18 yo
* Pregnancy or lactation
* Heavy smokers (>10 die)
* Conditions or diseases influencing periodontal healing
* Patients that cannot complete the 6 months follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Change in pocket closure % (0 - 100 % with higher percentage indicating better status) | [Time Frame: Baseline, 1 month, 3 months and 6 months after the completion of the therapy.]
  Percentage of pockets ≥ 5 mm that converted to ≤4 mm at the completion of NSPT

SECONDARY OUTCOMES:
Change in Full Mouth Plaque Score (FMPS%) (0 - 100 % with higher percentage indicating worse status) | [Time Frame: Baseline, 1 month, 3 months and 6 months after the completion of the therapy.]
  Percentage of full mouth plaque score considering 6 sited for each tooth.
Change in Probing Pocket Depth (PD) (0 - 15 mm with higher values indicating worse outcomes. | [Time Frame: Baseline, 1 month, 3 months and 6 months after the completion of the therapy.]
  The distance between the cementoenamel junction (CEJ) and the base of the pocket.
Change in Clinical Attachment Level (CAL) (0 - 15 mm with higher values indicating worse outcomes. | [Time Frame: Baseline, 1 month, 3 months and 6 months after the completion of the therapy.]
  The sum of Probing pocket depth (PD, mm) and Recession (Rec, mm)
Monetary cost for the treatment plan in € | [Time Frame: 1 month, 3 months and 6 months after the completion of the therapy.]
  Cost in € for the proposed treatment plan for patient at each re-evaluation timing based on the Italian Dental Association survey of charges for periodontal services for general dentists and periodontists.

CONTACTS AND LOCATIONS:
Locations (1):
- CIR Dental School, Turin, Italy

REFERENCES:
- [Derived] Baima G, Dabdoub S, Thumbigere-Math V, Ribaldone DG, Caviglia GP, Tenori L, Fantato L, Vignoli A, Romandini M, Ferrocino I, Aimetti M. Multi-Omics Signatures of Periodontitis and Periodontal Therapy on the Oral and Gut Microbiome. J Periodontal Res. 2025 Nov 27. doi: 10.1111/jre.70055. Online ahead of print. PMID 41307322
- [Derived] Baima G, Ferrocino I, Del Lupo V, Colonna E, Thumbigere-Math V, Caviglia GP, Franciosa I, Mariani GM, Romandini M, Ribaldone DG, Romano F, Aimetti M. Effect of Periodontitis and Periodontal Therapy on Oral and Gut Microbiota. J Dent Res. 2024 Apr;103(4):359-368. doi: 10.1177/00220345231222800. Epub 2024 Feb 16. PMID 38362600
- [Derived] Ferrarotti F, Baima G, Rendinelli M, Citterio F, Mariani GM, Mussano F, Romano F, Romandini M, Aimetti M. Pocket closure after repeated subgingival instrumentation: a stress test to the EFP guideline for stage III-IV periodontitis. Clin Oral Investig. 2023 Nov;27(11):6701-6708. doi: 10.1007/s00784-023-05279-6. Epub 2023 Sep 29. PMID 37773418